CLINICAL TRIAL: NCT04481113
Title: A Phase 1 Study of Abemaciclib and Niraparib as Neoadjuvant Therapy in Hormone Receptor Positive (HR+) HER2 Negative (HER2-) Breast Cancer
Brief Title: Abemaciclib and Niraparib Before Surgery for the Treatment of Hormone Receptor Positive HER2 Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry); GlaxoSmithKline (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alexandra Zimmer, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00021243; NCI-2020-03813 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00021243 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-04

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; HER2 Negative Breast Adenocarcinoma; Hormone Receptor Positive Breast Adenocarcinoma; Invasive Breast Carcinoma; Multifocal Breast Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Unilateral Breast Carcinoma
MeSH Terms: conditions — Unilateral Breast Neoplasms | interventions — abemaciclib; niraparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (abemaciclib, niraparib) (Experimental): Patients receive abemaciclib PO BID and niraparib PO QD. Treatment repeats every 28 days for up to 2-4 cycles in the absence of disease progression or unacceptable toxicity. Patients who complete 4 cycles undergo standard of care mastectomy or lumpectomy. Patients demonstrating progressive disease after only 2 cycles are switched to receive standard of care chemotherapy prior to undergoing mastectomy or lumpectomy.
  Interventions: Drug: Abemaciclib; Drug: Niraparib Tosylate Monohydrate

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY-2835219; LY2835219; Verzenio
Drug: Niraparib Tosylate Monohydrate — Given PO
  Other Names: Zejula

SUMMARY:
This phase I trial tests the side effects and best dose of abemaciclib and niraparib in treating patients with breast cancer that is positive for estrogen or progesterone receptors (hormone receptor positive [HR+]) and HER2 negative. Abemaciclib may stop the growth of tumor cells by blocking certain proteins called cyclin-dependent kinases, which are needed for cell growth. PARPs are proteins that help repair DNA mutations. PARP inhibitors, such as niraparib, can keep PARP from working so tumor cells can't repair themselves and grow. Giving abemaciclib and niraparib together before surgery may make the tumor smaller.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD) and/or recommended phase 2 dose of the combination of abemaciclib and niraparib tosylate monohydrate (niraparib).

II. To assess safety and tolerability of the combination of abemaciclib and niraparib in early stage HR+ breast cancer.

SECONDARY OBJECTIVES:

I. To determine clinical response to treatment. II. To determine pathologic response to treatment. III. To determine feasibility of combination as determined by no delay to standard of care breast surgery.

EXPLORATORY OBJECTIVE:

I. To assess occurrence of secondary myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) malignancy.

OUTLINE: This is a phase 1 dose-escalation study of abemaciclib in combination with niraparib followed by a dose-expansion study.

Patients receive abemaciclib orally (PO) twice daily (BID) and niraparib PO once daily (QD). Treatment repeats every 28 days for up to 2-4 cycles in the absence of disease progression or unacceptable toxicity. Patients who complete 4 cycles undergo standard of care mastectomy or lumpectomy. Patients demonstrating progressive disease after only 2 cycles are switched to receive standard of care chemotherapy prior to undergoing mastectomy or lumpectomy.

Patients are followed up at 30 days after date of surgery, every 3 months for the first 6 months, every 6 months for 2 years, then annually for up to 5 years from date of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Females (regardless of menopausal status), or males
* Biopsy proven estrogen receptor (ER) and/or progesterone receptor (PR) positive as defined as ER >= 1% and/or PR >= 1% by immunohistochemistry according to American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines for hormone receptor testing
* HER2 non-amplified per 2018 ASCO/CAP guidelines, defined as:

  * Immunohistochemistry (IHC) score 0/1+, or
  * IHC 2+ and in situ hybridization (ISH) non-amplified with a ratio of HER2 to CEP17 < 2.0, and if reported, average HER2 gene copy number < 4 signals/cells; or
  * ISH non-amplified with a ratio of HER2 to CEP17 < 2.0, and if reported, average HER2 gene copy number < 4 signals/cells
* Clinical T1-T3, any N, M0 invasive breast cancer, by American Joint Committee on Cancer (AJCC) 8th edition clinical staging with the goal being curative intent surgery to completely excise involved tumor in the breast and the draining lymph nodes
* Individuals with unilateral, multi-focal breast cancer (defined as more than one lesion of invasive breast cancer in the same breast separated from the dominant breast lesion by less than 5 cm of radiologically normal breast tissue) are eligible
* Participants must be planned for neoadjuvant chemotherapy
* Except for allowable endocrine therapy up to 4 weeks prior to study enrollment, participants must not have received prior anti-cancer therapy for the treatment of their breast cancer
* Participant must have disease that is amenable to biopsy, and agree to provide the required research biopsies at baseline, and 2 months after initiating study therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* The participant is able to swallow oral medications
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN). Participants with Gilbert's syndrome with a total bilirubin =< 2.0 times ULN and direct bilirubin within normal limits are permitted
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN
* If a participant is a cancer survivor, they have undergone potentially curative therapy for all prior malignancies, with no evidence of recurrence > 5 years
* Female participants of childbearing potential (FOCBP) must have a negative serum or high sensitive urine pregnancy test (per institutional standards) within 7 days prior to the start of study drugs
* FOCBP must agree to use highly-effective method(s) of contraception during the study and for 6 months after the last dose of study drugs
* FOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year without an alternative medical cause
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through at least 3 months after the last dose of study drugs
* Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment
* Participants receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy
* Participant must agree to not breastfeed during the study or for 30 days after the last dose of study treatment
* The participant must have normal BP or adequately treated and controlled hypertension (systolic BP <=140 mmHg and diastolic BP ≤90 mmHg).

Exclusion Criteria:

* Prior history of malignancy within 5 years except for successfully treated cervical carcinoma in situ, lobular carcinoma in situ of the breast, or non-melanoma skin cancer
* Inflammatory breast cancer defined as clinically significant erythema of the breast and/or documented dermal lymphatic invasion (not direct skin invasion by tumor or peau d'orange without erythema) is not eligible
* Participants that have undergone surgical axillary staging procedure prior to study entry

  * Fine needle aspiration (FNA) or core needle biopsy of axillary node is permitted
* Bilateral breast cancer, except for those tumors exhibiting similar biomarkers (grade, ER/PR, HER2)
* Clinical or radiographic evidence of metastatic disease

  * Isolated ipsilateral supraclavicular node involvement is permitted
  * A prior history of ductal breast carcinoma in situ (DCIS) treated with contralateral mastectomy and not receiving endocrine therapy is eligible
* Breast implants are contraindicated only if the implant precludes the required research biopsies or interferes with palpating the breast lesion
* Prior treatment for this cancer including surgery, radiation therapy, chemotherapy, biotherapy, hormonal therapy or investigational agent prior to study entry

  * Participants may have received up to 4 weeks of endocrine therapy prior to enrollment on trial
* Participants with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)
* Contraindication to undergoing breast and/or axillary lymph node biopsy
* Contraindication to undergoing surgical resection
* Prior therapy with a PARP inhibitor
* Prior therapy with a CDK 4/6 inhibitor
* The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [e.g., hepatitis B surface antigen positive]. Screening is not required for enrollment
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance < 30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea)
* Known history of pneumonitis or interstitial lung disease (ILD)
* Known history of deep vein thrombosis (DVT) or pulmonary embolism (PE)
* Participant must not have received a transfusion (platelets or red blood cells) =< 4 weeks prior to initiating protocol therapy. Exceptions may be made at the discretion of the investigator for the treatment of clinical complications such as bleeding. In these cases, protocol therapy may start >= 7 days after transfusion
* Participant must not have received colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior to initiating protocol therapy
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
* Resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, Fridericia's Correction Formula (QTcF) prolongation > 500 ms, electrolyte disturbances, etc.), or participants with congenital long QT syndrome
* Uncontrolled hypertension, or hypertension that cannot otherwise be clinically managed before initiating study therapy
* Psychiatric illness/social situations, or any condition that, in the opinion of the investigator, would: interfere with evaluation of study treatment or interpretation of participant safety or study results, or substantially increase risk of incurring adverse events (AEs), or compromise the ability of the patient to give written informed consent
* Participant must not have had major surgery =< 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects
* Hypersensitivity to any study agent, or its excipients, when administered alone
* Females who are pregnant or lactating
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) for the proposed combination | First dose of study agents to end of cycle 1 for dose-determining phase (each cycle is 28 days)
  Dose-limiting toxicities will specifically be reported for the DLT evaluation period using the MTD-evaluable population.
Incidence of adverse events (AEs) and serious AEs for the proposed combination | Up to 90 days from last dose of study agent (up to 7 months)
  Adverse events will be tabulated by the Medical Dictionary for Regulatory Activities (MedDRA version 21.1) preferred term and system organ class and a preferred term. The severity of the AEs will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 criteria. Descriptive statistics using the safety evaluable population will be used to report on all on-study AEs, grade 3-4 AEs, treatment-related AEs, grade 3-4 treatment-related AEs, serious adverse events (SAEs), treatment-related SAEs, and AEs leading to discontinuation per CTCAE v5.0. Grade 3-4 laboratory abnormalities will be summarized using worst grade NCI CTCAE v 5.0 criteria.

SECONDARY OUTCOMES:
Overall objective response rate (ORR) | From the date of first dose of study agents to 30 days post-surgery (up to 5 months)
  Overall response will be summarized descriptively. ORR will be estimated with 95% confidence interval (CI). The CI will be calculated based on the exact method for binomial distributions.
Clinical benefit rate (CBR) | From date of dose of study agents to 30 days post-surgery (up to 5 months)
  An estimate of CBR will be measured and reported with 95% exact CI. Participants who achieve a complete response (CR), partial response (PR), or stable disease (SD) for at least 6 months on the current protocol will be qualified as deriving benefit from therapy and will count towards the CBR measurement.
Rate of pathological complete response (pCR) | At time of surgical resection (up to 4 months)
  pCR will be tabulated as proportions and analyzed descriptively. Rate of delay to breast surgery will be summarized descriptively
Rate of residual cancer burden (RCB) 0-1 | At time of surgical resection (up to 4 months)
  RCB will be tabulated as proportions and analyzed descriptively. Rate of delay to breast surgery will be summarized descriptively
Rate of delay to breast surgery | From date of last dose of study drug to date of surgery (up to 4 months)
  Defined as proportion of participants with time-to-surgery > 90 days following completion of study therapy due to study-treatment related toxicity.

OTHER OUTCOMES:
Incidence of myelodysplastic syndrome/acute myeloid leukemia | Up to 5 years from the last dose of study drugs

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Zimmer, M.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States